CLINICAL TRIAL: NCT00122577
Title: Randomized Open Label Study Assessing the Antiviral Activity, Toxicity and Pharmacologic Interaction of Tenofovir DF/Atazanavir Enhanced With Low Dose of Ritonavir as Part of a Salvage Regimen in HIV Infected Patients With Multiple Treatment Failures (ANRS 107 Trial PUZZLE 2)
Brief Title: Efficacy and Safety of Tenofovir DF/Atazanavir Enhanced With Low Dose of Ritonavir in HIV-Infected Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Bristol-Myers Squibb (Industry); Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 107 Puzzle 2
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2005-07-28 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: HIV infections; Treatment Failure; tenofovir; atazanavir
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Atazanavir Sulfate; Ritonavir

INTERVENTIONS:
Drug: Tenofovir
Drug: Atazanavir
Drug: Ritonavir

SUMMARY:
This trial is aimed at studying the antiviral activity, toxicity and pharmacokinetic (PK) interactions of tenofovir DF and atazanavir enhanced with low dose of ritonavir given alone and then concomitantly as part of a salvage regimen to HIV patients with multiple failure, under conditions allowing to tease out the specific role of atazanavir combined with low dose of ritonavir.

DETAILED DESCRIPTION:
When licensed, new drugs are widely used in patients failing antiretroviral therapy, including patients with multiple failures. In such patients, having multi-resistant virus, the introduction of one new drug only in the salvage regimen will infrequently result in undetectable virus load in the plasma. Tenofovir DF and atazanavir appear promising because of their pharmacokinetic profile, activity, safety and resistance properties. In addition, pharmacokinetic data in healthy volunteers suggest that atazanavir could be optimized by adding ritonavir at low dose. Thus, one may speculate that atazanavir pharmacokinetic and antiviral activity could be optimized by adding ritonavir at low dose in patients exhibiting high rate of protease inhibitor mutations.

This protocol is aimed at studying the antiviral activity, toxicity and PK interactions, of tenofovir DF and atazanavir enhanced with low dose of ritonavir given alone and then concomitantly as part of a salvage regimen to patients with multiple failure, under conditions allowing to tease out the specific role of atazanavir combined with low dose of ritonavir.

EKG abnormalities (increased PR and QTc intervals) were observed in normal volunteers treated with atazanavir, therefore EKG safety monitoring will be performed on all subjects during this study

ELIGIBILITY:
Inclusion Criteria:

* Males and non pregnant females 18 years of age and older who have confirmed laboratory diagnosis of HIV infection and documented failure (plasma HIV RNA level over 10,000 copies/ml) to at least two protease inhibitors (ritonavir [RTV] must have been given at a dose over 400 mg twice a day (bid), in order to qualify for a protease inhibitor in this study) and one non-nucleoside reverse transcriptase inhibitor (NNRTI)
* Ongoing antiretroviral therapy at inclusion without change within the last month
* No threshold of CD4 cell count
* Patients naive of atazanavir and tenofovir DF

Exclusion Criteria:

* Cardiomyopathy
* QTc interval over 450 msec and pause length over 3 seconds on screening EKG
* Heart rate below 40 bpm
* Third degree heart block, and clinical symptoms potentially related to heart block
* Ongoing immunotherapy including IL2, interferon or HIV specific vaccine
* Ongoing opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-03; Study Completion 2004-07

PRIMARY OUTCOMES:
Change in plasma HIV RNA level and percentage of patients with undetectable HIV-RNA in plasma at Week 26

SECONDARY OUTCOMES:
Tolerance during the study
Changes in CD4+ counts at week 26
Emergence of drug-resistant viruses
Rate of virus decay in plasma in group 2 during the initial phase (14 days) of therapy according to baseline EC50 of atazanavir
Pharmacokinetic (PK) profile of atazanavir alone at day 14
Blood samples prior to drug administration (Cmin) and after drug administration on day 14 at +1h, +2h, +3h, +5h, +8h, and +24h in 10 patients of group 2
PK assessment on Week 6, of atazanavir, after 4 weeks of co-administration with tenofovir DF. (Blood samples prior to drug administration (Cmin) and after drug administration at +1h, +2h, +3h, +5h, +8h, and +24h in the same 10 patients of group 2)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Piketty, MD, Principal Investigator — Hopital Européen Georges Pompidou Paris, service d'immunologie clinique; Jean Pierre Aboulker, MD, Study Chair — Inserm SC10
Locations (1):
- Service d'Immunologie clinique Hopital Europeen Georges Pompidou, Paris, France

REFERENCES:
- [Result] Piketty C, Gerard L, Chazallon C, Calvez V, Clavel F, Taburet AM, Girard PM, Aboulker JP; ANRS 107 Puzzle 2 Study Group. Virological and immunological impact of non-nucleoside reverse transcriptase inhibitor withdrawal in HIV-infected patients with multiple treatment failures. AIDS. 2004 Jul 2;18(10):1469-71. doi: 10.1097/01.aids.0000131340.68666.21. PMID 15199325
- [Result] Taburet AM, Piketty C, Chazallon C, Vincent I, Gerard L, Calvez V, Clavel F, Aboulker JP, Girard PM. Interactions between atazanavir-ritonavir and tenofovir in heavily pretreated human immunodeficiency virus-infected patients. Antimicrob Agents Chemother. 2004 Jun;48(6):2091-6. doi: 10.1128/AAC.48.6.2091-2096.2004. PMID 15155205